CLINICAL TRIAL: NCT05541796
Title: Clinical Outcomes and Patient Satisfaction Following Implantation of Tecnis Synergy and Tecnis Symfony Intraocular Lens
Brief Title: Clinical Outcomes Following Implantation of Tecnis Synergy and Symfony Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George O. Waring IV (Other)
Collaborators: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor-Investigator, George O. Waring IV, Principal Investigator, Waring Vision Institute
Organization: Waring Vision Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVI/2022/01
Record Dates: First submitted 2022-08-30; First posted 2022-09-15 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cataract
Keywords: Cataract; Tecnis Synergy; Tecnis Symfony; presbyopia-correcting intraocular lens
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Intervention Model Description: Prospective, non-comparative, interventional, phase 4 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Contralateral implantation of Tecnis Synergy and Tecnis Symfony IOLs (Other): Non-comparative study involving contralateral implantation of Tecnis Synergy and Tecnis Symfony IOLs.
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens — Tecnis Symfony Optiblue (Johnson & Johnson Vision, Santa Ana, CA, Unites States) is a violet light filtering extended depth of focus IOL that provides a continuous range of clear vision at far and intermediate.
  Tecnis Synergy™ IOL (Johnson & Johnson Vision, Santa Ana, CA, Unites States) is another latest United States Food and Drug Administration (USFDA) approved IOL, designed to provide good acuity at far through near distances, reducing the need for spectacles.

SUMMARY:
Tecnis Symfony Optiblue (Johnson & Johnson Vision, Santa Ana, CA, Unites States) is a violet light filtering extended depth of focus intraocular lens (IOL) that provides a continuous range of clear vision at far and intermediate. Tecnis Synergy™ IOL (Johnson & Johnson Vision, Santa Ana, CA, Unites States) is another latest United States Food and Drug Administration (USFDA) approved IOL, designed to provide good acuity at far through near distances, reducing the need for spectacles. These IOLs are approved/licensed for use and are not investigational. The present study intends to evaluate the clinical outcomes and patient satisfaction following contralateral implantation of Tecnis Synergy and Symfony Optiblue in cataract patients. The investigator hypothesizes that the contralateral implantation of these two lenses will allow a good proportion of patients to be spectacle independent at distance, intermediate, and near. The findings of this study may help the surgeons make better decisions on the choice of IOL in the future.

DETAILED DESCRIPTION:
Presbyopia-correcting intraocular lenses (IOLs), including multifocal and extended depth of focus (EDOF) IOLs, have revolutionized the field of refractive cataract surgery by providing good vision at multiple distances and spectacle independence. While multifocal IOLs provide good visual acuity at various distances, increased incidence of photic phenomena (haloes, glare, starbursts, etc.) associated with multifocal IOLs is a cause of dissatisfaction among patients. EDOF IOLs, on the other hand, are based on the principle of creating a single-elongated focal point to enhance the depth-of-focus (DOF) and eliminate the overlapping of near and far images caused by traditional multifocal IOLs, thus minimizing the halo effect.

Recent developments in IOL technologies focus on finding the best compromise between the range of visual rehabilitation and the induction of postoperative photic phenomena and contrast sensitivity reduction. One of these developments is the Tecnis Synergy™ IOL, which combines an EDOF profile with a multifocal diffractive design, to obtain continuous high-contrast vision from far through near, even in low-lighting conditions (Tecnis Synergy, Johnson & Johnson Vision, Santa Ana, CA, Unites States) without the visual gaps caused by the trifocal technology. Preliminary data with Tecnis Synergy IOLs in European populations are quite encouraging. In some cases, a combination of two different IOLs has been implanted to capitalize on the strengths and mitigate the weaknesses of each. Thus, the present study aims to evaluate the clinical outcomes and patient satisfaction following implantation of a combination of Tecnis Synergy and Tecnis Symfony OptiBlue IOLs in a US-based population of cataract surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Requiring bilateral cataract surgery, wish to achieve spectacle independence.
* Are suitable candidates for Tecnis Synergy and Tecnis Symfony IOLs
* Have predicted postoperative astigmatism ≤ 0.75 D
* Willing to provide written informed consent and adhere to study requirements

Exclusion Criteria:

* History of ocular surgery, including laser refractive surgery
* History of ocular trauma
* Patients planning for any concomitant ocular procedure at the time of cataract surgery (including MIGS) other than incisional correction of astigmatism as the time of surgery
* Ocular comorbidities including glaucoma, macular degeneration, corneal scars, or any other condition that might limit the ability to achieve 20/20 visual acuity.
* Unwillingness to provide written informed consent,
* Disability to understand and/or fill the patient questionnaire,
* Pregnancy or lactation.
* Any patient who meets enrollment criteria but subsequently experiences an intraoperative complication or does not undergo surgery with implantation of the intended pair of IOLs will also be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Binocular distance-corrected intermediate visual acuity under photopic conditions. | Postoperative 6 months
  Mean logMAR binocular distance-corrected intermediate visual acuity (DCIVA, 66 cm).
Binocular distance-corrected near visual acuity under photopic conditions. | Postoperative 6 months
  Mean logMAR binocular distance-corrected near visual acuity (DCNVA, 40 cm).
Binocular distance-corrected very near visual acuity under photopic conditions. | Postoperative 6 months
  Mean logMAR binocular distance-corrected very near visual acuity (DCVNVA, 33 cm).

SECONDARY OUTCOMES:
Binocular uncorrected intermediate visual acuity under photopic conditions | Postoperative 6 months
  Mean logMAR binocular uncorrected intermediate visual acuity measured at 66 cm
Binocular uncorrected near visual acuity under photopic conditions | Postoperative 6 months
  Mean logMAR binocular uncorrected near visual acuity measured at 40 cm
Binocular uncorrected very near visual acuity under photopic conditions | Postoperative 6 months
  Mean logMAR binocular uncorrected very near visual acuity measured at 33 cm
Binocular uncorrected distance visual acuity under photopic conditions | Postoperative 6 months
  Mean logMAR binocular uncorrected distance visual acuity
Subjective assessment of patient satisfaction and other patient-reported outcomes using visual symptoms questionnaire (PRVSQ) | Postoperative 6 months
  Subjective assessment of patient satisfaction with the surgery and other patient-reported outcomes using a patient-reported visual symptoms questionnaire (PRVSQ)
Subjective assessment of patient satisfaction and other patient-reported outcomes using spectacle independence questionnaire (PRSIQ) | Postoperative 6 months
  Subjective assessment of patient satisfaction with the surgery and other patient-reported outcomes using a patient-reported spectacle independence questionnaire (PRSIQ)

OTHER OUTCOMES:
Binocular distance-corrected intermediate visual acuity under mesopic conditions | Postoperative 6 months
  Binocular mean logMAR distance-corrected intermediate visual acuity (DCIVA, 66 cm)
Binocular distance-corrected near visual acuity under mesopic conditions | Postoperative 6 months
  Binocular mean logMAR distance-corrected near visual acuity (DCNVA, 40 cm)
Binocular distance-corrected very near visual acuity under mesopic conditions | Postoperative 6 months
  Binocular mean logMAR distance-corrected very near visual acuity (DCVNVA, 33 cm)
Binocular uncorrected distance visual acuity under mesopic conditions | Postoperative 6 months
  Binocular mean logMAR uncorrected distance visual acuity
Binocular uncorrected intermediate visual acuity under mesopic conditions | Postoperative 6 months
  Binocular mean logMAR uncorrected intermediate visual acuity (UIVA, 66 cm)
Binocular uncorrected near visual acuity under mesopic conditions | Postoperative 6 months
  Binocular mean logMAR uncorrected near visual acuity (UNVA, 40 cm)
Binocular uncorrected very near visual acuity under mesopic conditions | Postoperative 6 months
  Binocular mean logMAR uncorrected very near visual acuity (UVNVA, 33 cm)

CONTACTS AND LOCATIONS:
Overall Officials: George O Waring IV, MD FACS, Principal Investigator — Waring Vision Institute
Locations (1):
- Waring Vision Institute, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No